CLINICAL TRIAL: NCT02098525
Title: Clinical Outcomes of Cryptococcal Meningitis Among HIV-infected Patients in the Era of Antiretroviral Therapy
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Prof., Mahidol University
Other Study IDs: HIVCM-01
Record Dates: First submitted 2014-03-18; First posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Cryptococcal Meningitis; HIV/AIDS
Keywords: Cryptococcal meningitis; HIV/AIDS; Antiretroviral therapy; Prognosis; Thailand
MeSH Terms: conditions — Meningitis, Cryptococcal; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV associated CM patients: The study population is all adult HIV positive patients with CM at Ramathibodi Hospital.

SUMMARY:
Cryptococcal meningitis is one of the most common central nervous system infections among HIV-infected patients. The outcome is generally severe. This study aims to determine long-term survival rate among HIV-infected CM patients in the era of antiretroviral therapy (ART). The secondary objectives are to clarify outcomes of CM and determine prognostic factors.

DETAILED DESCRIPTION:
Study site:

The study are conducted at the Division of Infectious Diseases, Department of Medicine, Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand.

Sample size calculation:

The sample size is obtained by using EPI Info program. Anticipated population proportion P which will be the major outcome of CM, the survival rate was 63% in Thailand (Chottanapund S, Singhasivanon P, Kaewkungwal J, Chamroonswasdi K, Manosuthi W. Survival time of HIV-infected patients with cryptococcal meningitis. J Med Assoc Thai. 2007 Oct;90(10):2104-11. PubMed PMID: 18041430). At the effect size of 80%, confidence level at 95% (P = 0.05), deviation error of allowanced of 5% and 210 expects HIV infected patients with CM during study period at Ramathibodi Hospital, the estimated sample size is 132 cases.

Outcome measurement:

Death case: Death case is CM patient who died for any reason during the period of follow-up.

Survival case: Survival case is CM patient who did not die during the period of follow-up.

Relapse case: This refers to a patient who developed a new episode of CM after clinical manifestations had disappeared and CSF culture had become negative, and confirmed by positive CSF culture for Cryptococcus neoformans.

IRIS case: This refers to a patient who developed a new episode of clinical meningitis after clinical manifestations stemming from a previous episode of CM had disappeared and the patient had been started ART, and defined as negative CSF culture for Cryptococcus neoformans. Alternative etiology which presents symptoms similar to CM must be ruled out.

Clinical outcome parameters:

Short-term outcome: Short-term outcome is defined as the outcome that happened within 1 year of follow up period.

Long-term outcome: Long-term outcome is defined as all outcomes that happened after 1 year of follow up period.

Margin period to evaluate the blood findings at AmB induction therapy initiation is defined as within 3 months from the exact date of AmB induction therapy initiation.

Margin period to evaluate the parameters at AmB induction therapy completion is defined as within 7 days from the exact date of AmB induction therapy completion.

Margin period to evaluate the CSF findings at ART initiation is defined as within 1 month from the exact date of ART initiation.

Margin period to evaluate the blood findings at ART initiation is defined as from 3 months before to 1 month after the exact date of ART initiation.

Margin period to evaluate the parameters at secondary FLCZ prophylaxis completion is defined as within 3 months from the exact date of secondary FLCZ prophylaxis completion.

Research methodology:

The medical records of those diagnosed with HIV associated CM is retrieved from the medical record department in Ramathibodi Hospital. Then the inclusion and exclusion criteria are checked. We review at least 132 cases. The information from the medical records which pass the criteria is extracted and transferred to the case report form. Then data entry is carried out with coding and verified.

Statistical analysis:

The data will be computed by means of the descriptive statistical methods as the following values: frequency distribution, proportion, rate, median and range. To compare demographic and clinical characteristics, we will use chi-square tests or Fisher's exact tests for categorical variables and student's t tests or Mann-Whitney U tests for continuous variables. Cox's proportional hazards model and Kaplan-Meier survival analysis will be used to evaluate factors associated with outcomes. Hazard ratio, odds ratio and 95% CI will be calculated and used as a measure of the strength of the association between the outcome variables and their predictors. A two-tailed alpha level of 0.05 will be used to determine statistical significance. Statistical analyses will be performed with the statistical program, SPSS.

Ethical committee approval:

As a retrospective study, we review patients' medical records only. No patient are directly involved in this study and therefore no informed consent is obtained. The proposal is reviewed by the Ethical Committee of the Faculty of Tropical Medicine, Mahidol University, for clearance. Data collection was started after the protocol is ethically approved.

Confidentiality:

The names or any clues leading to the identification of the patients are not be recorded in CRF (case record form). Only code numbers are recorded in CRF. The information of patient's identification and code number are kept separately. The results are presented as medical data with no personal identifying information. Authorized person helps to collect data.

Research funds:

Funding for the study is provided by the Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients diagnosed by positive results of 2 different ELISA tests, 1 ELISA test accompanied with 1 HIV-PCR test, or 1 ELISA test accompanied with 1 Western blot test, whose age was more than 15 years old.
* Newly diagnosed CM during the study period defined by positive culture, positive Indian ink or positive latex agglutination test on CSF with typical symptoms at Ramathibodi Hospital.

Exclusion Criteria:

* Patients who had other known CNS co-infection or other significant concurrent CNS diseases which might influence on outcome of CM.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is all adult HIV positive patients with CM at Ramathibodi Hospital, Mahidol University.
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Long-term survival rate of CM | Up to 12 years. Cases will be censored at the date of last visit if they are lost to follow up or referred to another hospital, and will be censored at the date of death.
  To describe long-term survival rate of CM among adult HIV-infected patients in the era of ART.

SECONDARY OUTCOMES:
Risk factors of short-term and long-term mortality of CM | Up to 12 years. Cases will be censored at the date of last visit if they are lost to follow up or referred to another hospital, and will be censored at the date of death.
  To identify risk factors of short-term and long-term mortality of CM.

CONTACTS AND LOCATIONS:
Overall Officials: Taiichiro Kobayashi, Dr, Principal Investigator — Mahidol University; Punnee Pitisuttithum, Prof., Study Director — Mahidol University; Weerawat Manosuthi, Dr., Study Chair — Bamrasnaradura infectious disease hospital
Locations (1):
- Division of Infectious Diseases, Department of Medicine, Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Bangkok, Thailand